CLINICAL TRIAL: NCT00968162
Title: Toward a Less Toxic Yet Highly Effective Conditioning Regimen in Allogeneic Hematopoietic Stem Cell Transplantation for Children and Adolescents With Severe Sickle Cell Disease: A Pilot Study
Brief Title: Sickle Cell Disease Conditioning for Bone Marrow Transplant
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, John Horan, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00011048; BMT for SCD (Other: Other)
Record Dates: First submitted 2009-08-11; First posted 2009-08-28 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Bone Marrow Transplantation; Sickle Cell Disease
Keywords: Bone Marrow Transplant; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose de-escalation (Experimental)
  Interventions: Drug: fludarabine

INTERVENTIONS:
Drug: fludarabine — Conduct a pilot trial using a transplant protocol, in which the standard busulfan, cyclophosphamide and anti-thymocyte globulin conditioning regimen is modified by adding fludarabine, a highly immunosuppressive agent, in order to determine the feasibility of reducing the total dose of cyclophosphamide from its present standard of 200 mg/kg to 90 mg/kg and of busulfan from its present standard of 12.8 mg/kg (IV) to 6.4 mg/kg, using a four step dose de-escalation schema.

SUMMARY:
Most bone marrow transplants for children with sickle cell disease are performed using high doses of two chemotherapy agents: busulfan and cyclophosphamide for the pre-transplant conditioning. This approach produces cure in most cases (approximately 95%). It, however, has serious side effects, including seizures and infertility. The primary goal of this study is to determine how much we can lower the dosages of busulfan and cyclophosphamide by incorporating fludarabine, a safer chemotherapy agent, into conditioning. The secondary goal is to develop a better understanding of how bone marrow transplants cause neurologic problems like seizures.

DETAILED DESCRIPTION:
Many children with sickle cell disease are severely affected by acute complications, especially stroke, recurrent and debilitating pain, or recurrent acute chest syndrome. As they become adolescents and young adults, patients with sickle cell disease often develop chronic problems, including renal disease, chronic lung disease and pulmonary hypertension. For children who have an HLA matched related donor, a hematopoietic stem cell transplant (HSCT), using bone marrow or cord blood is an effective cure; using the standard approach, which relies on high doses of busulfan (BU) and cyclophosphamide (CY) as well as anti-thymocyte globulin (ATG) for pre-transplant conditioning, the probability of event free survival is now approximately 95%. The standard approach, however, is frequently complicated by acute and often severe neurological events, such as seizure and encephalopathy, as well as hypogonadism. Circumstantial evidence suggests that sickle cell patients are predisposed to transplant related neurological toxicities by disease related cerebrovascular injury, and that the transplant process aggravates this injury, causing cerebral ischemia and, in turn, neurological toxicity. The high dose chemotherapy, which has been shown to induce endothelial injury, appears to be an important contributing factor. The role of high dose chemotherapy in transplant related neurotoxicity needs to be more firmly established. The role of high dose alkylating agents in gonadal injury has been well established. Fludarabine, a non-vasculopathic, non-gonadotoxic agent, amplifies the engraftment promoting effects of Cy; in an effort to lessen the incidence of transplant related neurotoxicity and gonadotoxicity, we will conduct a pilot study in which fludarabine is added to BuCyATG for conditioning, and the dose of Bu and Cy are reduced using a stepwise de-escalation schema. This study will serve as a forerunner to larger trial designed to test the safety and efficacy of a reduced toxicity BuFluCyATG regimen. Central Hypothesis: A safer approach to hematopoietic stem cell transplantation (HSCT) can be developed for children with sickle cell disease without compromising efficacy. Specific Aims: 1) To begin to develop a reduced dose busulfan and cyclophosphamide based conditioning regimen for children with sickle cell disease that still achieves sustained engraftment at least 90% of the time, by conducting a pilot trial, in which the standard busulfan, cyclophosphamide and anti-thymocyte globulin conditioning regimen is modified by adding fludarabine, a non-vasculopathic and non-gonadotoxic, yet highly immunosuppressive agent, in order to determine the feasibility of reducing the total dose of cyclophosphamide from its present standard of 200 mg/kg to 90 mg/kg and the busulfan from its present standard of 12.8 mg/kg (IV) to 6.4 mg/kg, using a four step dose de-escalation schema.. 2) a) To begin to assess the vascular, and more specifically, the cerebrovascular effects of pre-transplant, high-dose busulfan and cyclophosphamide in children with sickle cell disease by obtaining preliminary estimates of longitudinal changes in the blood levels biomarkers of endothelial dysfunction and inflammation (endothelin-1, von Willebrand factor antigen, C-reactive protein, Il-8 thrombin-antithrombin (TAT) complexes) and in the changes in two MRI biomarkers-cortical thickness measurement and diffusion tensor imaging.. b) To begin to assess the long-term effects of replacing sickle erythrocytes with normal erythrocytes (by HSCT) on the vasculature and cerebrovasculature, using the same tests. These estimates will help us to calculate a sample size and refine our testing for the second study.

ELIGIBILITY:
Inclusion Criteria:

1. Up to and including the age of 18 years at time of admission for transplant
2. Hemoglobin SS, or hemoglobin S0 thalassemia
3. HLA-identical sibling donor (any age) available without HgbSS, SC or S0 thalassemia. As an alternative, HLA identical sibling umbilical cord blood can be used as long as the unit has a pre-cryopreservation TNC dose of greater than 5.0 x 107 TNC/kg recipient weight.
4. Clinically severe SCD, defined by one of the following:

   1. Previous clinical stroke, as evidenced by a neurological deficit lasting longer than 24 hours, which is accompanied by radiographic evidence of ischemic brain injury and cerebral vasculopathy.
   2. Asymptomatic cerebrovascular disease, as evidenced by one the following:

   (i)Progressive silent cerebral infarction, as evidenced by serial MRI scans that demonstrate the development of a succession of lesions (at least two temporally discreet lesions, each measuring at least 3 mm in greatest dimension on the most recent scan) or the enlargement of a single lesion, initially measuring at least 3 mm). Lesions must be visible on T2-weighted MRI sequences.

   (ii) Cerebral arteriopathy, as evidenced by abnormal TCD testing (confirmed elevated velocities in any single vessel of TAMMV > 200 cm/sec for non-imaging TCD or TAMX > 185 cm/sec for imaging TCD) or by significant vasculopathy on MRA (greater than 50% stenosis of > 2 arterial segments or complete occlusion of any single arterial segment).

   (c) Frequent (≥ 3 per year for preceding 2 years) painful vaso-occlusive episodes (defined as episode lasting ≥ 4 hours and requiring hospitalization or outpatient treatment with parenteral opioids). If patient is on hydroxyurea and its use has been associated with a decrease in the frequency of episodes, the frequency should be gauged from the 2 years prior to the start of this drug.

   (d) Recurrent (≥ 3 in lifetime) acute chest syndrome events that have necessitated erythrocyte transfusion therapy.

   (e) Any combination of ≥ 3 acute chest syndrome episodes and vaso-occlusive pain episodes (defined as above) yearly for 3 years. If patient is on hydroxyurea and its use has been associated with a decrease in the frequency of episodes, the frequency should be gauged from the 3 years prior to the start of this drug.
5. Must have been evaluated and adequately counseled regarding treatment options for severe sickle cell disease by a pediatric hematologist.

Exclusion Criteria:

1. Biopsy proven chronic active hepatitis, portal fibrosis (greater than score I), or cirrhosis, or serologic evidence of active hepatitis.
2. SCD chronic lung disease stage III (see appendix 1).
3. Severe renal dysfunction defined as < 50% of predicted normal GFR for age.
4. Severe cardiac dysfunction defined as shortening fraction < 25%.
5. Severe residual neurologic impairment other than hemiplegia alone, defined as full-scale IQ 70, quadriplegia or paraplegia, inability to ambulate, inability to communicate without assistive device, or any impairment resulting in decline of Lansky performance score to < 70%.
6. CNS event occurring within 6 months prior to transplant.
7. Karnofsky or Lansky functional performance score < 70%.
8. Confirmed HIV seropositivity.
9. Patient with unspecified chronic toxicity serious enough to detrimentally affect the patient's capacity to tolerate bone marrow transplantation.
10. Patient or patient's guardian(s) unable to understand the nature and risks inherent in the BMT process.
11. History of lack of compliance with medical care that would jeopardize transplant course.
12. Donor who for psychological, physiologic, or medical reasons is unable to tolerate a bone marrow harvest or receive general anesthesia.
13. Donor is HIV infected.
14. Donor is pregnant.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2009-02; Primary Completion 2014-03 (Actual); Study Completion 2016-01-11 (Actual)

PRIMARY OUTCOMES:
Modify the standard dose of busulfan, cyclophosphamide and anti-thymocyte globulin conditioning regimen by adding fludarabine in order to determine the feasibility of reducing the total dose of cyclophosphamide from its present standard of 200 mg/kg. | 1 year after last patient enrolled

SECONDARY OUTCOMES:
To gain insight into the processes that give rise to neurologic problems following bone marrow transplantation and to develop surrogate outcomes. | 1 year after last patient enrolled

CONTACTS AND LOCATIONS:
Overall Officials: John Horan, MD, Principal Investigator — Emory University
Locations (10):
- United States (10):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Research Institute Inc., St. Petersburg, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Tulane University, New Orleans, Louisiana
  - Wayne State University, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Montefiore Medical Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - University of Texas Southwestern, Dallas, Texas